CLINICAL TRIAL: NCT05232032
Title: Pharmaco-Neuroimaging Studies of Approach/Avoidance Behaviors and Post-Mortem Studies: Study 1.1. (Pharmacological Manipulation)
Brief Title: Pharmaco-Neuroimaging Studies of Approach/Avoidance Behaviors and Post-Mortem Studies: Pharmacological Manipulation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Massachusetts General Hospital (Other); Massachusetts Institute of Technology (Other); University of Washington (Other); Brown University (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Professor, Department of Psychiatry, Harvard Medical School, McLean Hospital, McLean Hospital, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024P002715; 5P50MH119467-02 (NIH)
Record Dates: First submitted 2022-02-01; First posted 2022-02-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Depressive Disorder, Major; Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Participants with MDD or an anxiety disorder receiving the nociceptin receptor antagonist (Experimental): After a diagnostic interview (determining the presence of MDD or an anxiety disorder) and collection of blood for Orphanin FQ/Nociceptin assays, participants will receive the nociceptin receptor antagonist. Participants will then complete an approach/avoidance task. Functional magnetic resonance imagining (fMRI) will begin 2 hours after the nociceptin receptor antagonist is administered.
  Interventions: Drug: Nociceptin Receptor Antagonist; Device: Aversive stimuli
- Participants with MDD or an anxiety disorder receiving the placebo (Placebo Comparator): After a diagnostic interview (determining the presence of MDD or an anxiety disorder) and collection of blood for Orphanin FQ/Nociceptin assays, participants will receive the placebo. Participants will then complete an approach/avoidance task. fMRI will begin 2 hours after the placebo is administered.
  Interventions: Device: Aversive stimuli
- Healthy controls receiving the nociceptin receptor antagonist (Experimental): After a diagnostic interview (determining healthy control status) and collection of blood for Orphanin FQ/Nociceptin assays, participants will receive a nociceptin receptor antagonist. Participants will then complete an approach/avoidance task. fMRI will begin 2 hours after the nociceptin receptor antagonist is administered.
  Interventions: Drug: Nociceptin Receptor Antagonist; Device: Aversive stimuli
- Healthy controls receiving the placebo (Placebo Comparator): After a diagnostic interview (determining healthy control status) and collection of blood for Orphanin FQ/Nociceptin assays, participants will receive the placebo. Participants will then complete an approach/avoidance task. fMRI will begin 2 hours after the placebo is administered.
  Interventions: Device: Aversive stimuli

INTERVENTIONS:
Drug: Nociceptin Receptor Antagonist — Participants in the experimental arms will receive 40 mg of the nociceptin receptor antagonist. Peak concentrations are achieved 2-4 hours post-administration.
  Other Names: BTRX-246040
  Arms: Healthy controls receiving the nociceptin receptor antagonist; Participants with MDD or an anxiety disorder receiving the nociceptin receptor antagonist
Device: Aversive stimuli — As part of the approach/avoidance task, electrotactile stimulation will be used. The aversive stimulus is delivered in the form of a mild half-second stimulation to the ankle, calibrated to a subjective threshold that is uncomfortable but not painful. This stimulation is delivered by Digitimer DS8R Constant Current Stimulator (Digitimer North America, LLC. Ft. Lauderdale, FL). Its previous model, DS71, has been safely implemented in studies within Massachusetts General Hospital (Milad et al., 2013).

SUMMARY:
The study will investigate whether a nociceptin receptor antagonist will normalize neural and behavioral processes of approach/avoidance decision-making in unmedicated individuals with major depressive disorder (MDD) and anxiety disorders. More specifically, the study aims to investigate dysregulation within (1) corticostriatal-midbrain circuitry and (2) nociceptin/orphanin FQ peptide and the nociceptin receptor (NOPR).

ELIGIBILITY:
Inclusion criteria for MDD/anxiety disorder group:

* DSM-5 diagnostic criteria for MDD, Generalized Anxiety Disorder, Social Phobia, Panic Disorder, Post Traumatic Stress (diagnosed using the SCID-5)
* Written informed consent
* For MDD subjects, a baseline Hamilton Depression Rating Scale score > 16 (17-item version)
* Right-handed
* Has a smartphone (iPhone or Android) (needed for Ecological Momentary Assessment)
* Absence of any psychotropic medications for at least 2 weeks (6 weeks for fluoxetine, 6 months for neuroleptics, 2 weeks for benzodiazepines, 2 weeks for any other antidepressants)

Inclusion criteria for healthy controls:

* Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse), as assessed by subject history and a structured clinical interview (diagnosed using the SCID-5)
* Written informed consent
* Right-handed
* Absence of any medications for at least 3 weeks
* Has a smartphone (iPhone or Android) (needed for Ecological Momentary Assessment)

Exclusion criteria for all participants:

* Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician
* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder
* History or current diagnosis of any of the following DSM-IV psychiatric illnesses: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, obsessive-compulsive disorder, patients with mood congruent or mood incongruent psychotic features, substance dependence, substance abuse within the last 12 months (with the exception of cocaine or stimulant abuse; which will lead to exclusion)
* History of cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine)
* History of use of dopaminergic drugs (including methylphenidate)
* History or current diagnosis of dementia
* Patients with mood congruent or mood incongruent psychotic features
* Current use of other psychotropic drugs
* Clinical or laboratory evidence of hypothyroidism
* Patients with a lifetime history of electroconvulsive therapy
* Failure to meet standard magnetic resonance imaging safety requirements
* Abnormal ECG and lab results
* History of seizure disorder or currently on anticonvulsants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (SCID-5) | Baseline
  Diagnostic assessment
Magnetic Resonance Imagining | Within 30 days of the clinical interview
  Both structural and functional brain images
Approach/Avoidance Task | During the MRI scan
  A novel behavioral task assessing approach/avoidance decision-making
Orphanin FQ/Nociceptin assays (using blood samples) | On the day of the MRI scan
  Measure of Orphanin FQ/Nociceptin

SECONDARY OUTCOMES:
Beck Depression Inventory-II | Baseline, 6-month follow-up, 12-month follow-up
  21-item measure of depression severity; scores range from 0 to 63; higher scores indicate higher depression severity
Hamilton Rating Scale for Depression | Baseline, 6-month follow-up, 12-month follow-up
  17-item measure of depression severity; scores range from 0 to 34; higher scores indicate higher depression severity
Perceived Stress Scale | Baseline, 6-month follow-up, 12-month follow-up
  14-item measure of stress appraisal; scores range from 0 to 56; higher scores indicate higher perceived stress
Snaith Hamilton Pleasure Scale | Baseline, 6-month follow-up, 12-month follow-up
  14-item measure of anhedonia; scores range from 14 to 56; higher scores indicate higher anhedonia
Medical Outcome Survey- Short Form | Baseline, 6-month follow-up, 12-month follow-up
  36-item measure of physical and social functioning; score range from 36 to 149; higher scores indicate higher physical and social functioning
Quality of Life Enjoyment and Satisfaction Questionnaire | Baseline, 6-month follow-up, 12-month follow-up
  16-item measure of satisfaction and enjoyment across domains (e.g., work, interpersonal); scores range from 16 to 80; higher scores indicate higher life enjoyment and satisfaction
Temporal Experience of Pleasure Scale | Baseline, 6-month follow-up, 12-month follow-up
  24-item measure of anticipatory and consummatory pleasure; scores range from 24 to 144; higher scores indicate higher anticipatory/consummatory pleasure
Life Events and Difficulties Schedule | Baseline, 6-month follow-up, 12-month follow-up
  Measure of acute events, difficulties, stressors
Longitudinal Interval Follow-Up Evaluation (LIFE) (Keller et al., 1987) | 6-month follow-up, 12-month follow-up
  Retrospectively assesses different DSM-5 disorders, social and occupational functioning, and life satisfaction over the past 6 months
Columbia-Suicide Severity Rating Scale | Baseline, 6-month follow-up, 12-month follow-up
  Suicide assessment

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- Mclean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Through the Conte Center website, we will share de-identified data and tools with the scientific community (e.g., code developed by the Computational Modeling Core). In close collaboration with NIMH, we will develop a certification similar to the "NIMH Data Archive Data Use Certification" currently used by NIMH.
  Through the National Database for Clinical Trials Related to Mental Illness, we will share five principal human datasets generated within the Conte Center: (1) Clinical rating scales and self-report scales of affect, mood, symptoms and functioning; (2) Behavioral performance during approach-avoidance tasks; (3) Electrophysiological data; (4) Functional magnetic resonance imaging data; and (5) Hormonal (cortisol) responses.
  Through ClinicalTrials.gov, we will share the primary and secondary outcomes.